CLINICAL TRIAL: NCT02358824
Title: A Phase I Clinical Trial to Compare the Pharmacokinetics and Safety of CKD-828(Telmisartan 80mg/S-amlodipine 5mg Combination Tablet) to Coadministration of Telmisartan 80mg and S-amlodipine 5mg in Healthy Male Volunteers
Brief Title: CKD-828 (80/5mg) Pharmacokinetic Study
Acronym: CKD-828
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 130BE15002
Record Dates: First submitted 2015-02-04; First posted 2015-02-09 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Hypertension
Keywords: Hypertension; CKD-828; Telmisartan; S-amlodipine; Pharmacokinetic
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; levamlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CKD-828(Fixed Dose Combination) (Experimental): FDC tablet consisting of Telmisartan 80mg/S-Amlodipine 5mg
  Interventions: Drug: CKD-828
- Combination Therapy (Active Comparator): Coadministration of Telmisartan 80mg and S-amlodipine 5mg
  Interventions: Drug: Telmisartan; Drug: S-amlodipine

INTERVENTIONS:
Drug: CKD-828 — Telmisartan 80mg /S-Amlodipine 5mg(FDC) Tablet, Oral, Once Daily
  (1arm:2period and 4period, 2arm:1period and 3period)
  Other Names: Telminuvo
  Arms: CKD-828(Fixed Dose Combination)
Drug: Telmisartan — - Telmisartan 80mg tablet, Oral, Once Daily (Combination Therapy with S-amlodipine)
  (1arm:1period and 3period, 2arm: 2period and 4period)
  Other Names: Micardis
  Arms: Combination Therapy
Drug: S-amlodipine — - S-amlodipine 5mg tablet, Oral, Once Daily (combination Therapy with Telmisartan)
  (1arm:1period and 3period, 2arm: 2period and 4period)
  Other Names: Anydipine s
  Arms: Combination Therapy

SUMMARY:
A randomized, open-label, single-dose, four-period, two-way, crossover study,

DETAILED DESCRIPTION:
A randomized, open-label, single-dose, four-period, two-way, crossover study to compare the pharmacokinetics and safety CKD-828 (Fixed Dose Combination Tablet) to coadministration telmisartan and s-amlodipine in health volunteers.

ELIGIBILITY:
Inclusion Criteria:

* A healthy volunteer over 20 years old
* More than 50kg and within 20% of ideal body weight
* No any congenital or chronic diseases and medical symptom
* Appropriate for the study from examination(laboratory test, ECG etc.) within 4weeks prior to the first IP administration
* Signed the informed consent form prior to the study participation.

Exclusion Criteria:

* History of relevant hypersensitivity against drug
* Clinical significant disease or medical history (ex. hepato/cholangio, cardio, endo, hemato, onco, CNS etc.)
* Active liver disease or abnormal laboratory result (AST or ALT or Total bilirubin > 1.5*ULN)
* SBP <90mmHg or SBP >150mmHg
* DBP <50mmHg or DBP >100mmHg
* Creatinine clearance <80mL/min
* A Disease(ex.inflammatory intestinal disease, gastric or duodenal ulcer ,hepatic disease history , gastro-intestinal surgery except for appendectomy)that may influence on the absorption, distribution, metabolism and excretion of the drug
* The evidence of severe attack or acute disease or surgical intervention within 28 days prior to the first IP administration.
* A drug abuse or a heavy caffeine consumer (more than 5 cups per a day) or regular alcohol consumer(more than 21 units/week) or a heavy smoker(more than 10 cigarettes per a day)
* Taking ETC medicine or oriental medicine within 14days or Taking OTC medicine within 7days prior to the first IP administration
* Abnormal diet(Especially, grapefruit juice within 7 days prior to the first IP administration) that may influence on the absorption, distribution, metabolism and excretion of the drug

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-02; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Cmax after administration of CKD-828(Fixed Dose Combination) tablet and coadministration of corresponding dose of telmisartan and s-amlodipine. | up to 144 hours post dose
AUClast after administration of CKD-828(Fixed Dose Combination) tablet and coadministration of corresponding dose of telmisartan and s-amlodipine. | up to 144 hours post dose

SECONDARY OUTCOMES:
Tmax after administration of CKD-828(Fixed Dose Combination) tablet and coadministration of corresponding dose of telmisartan and s-amlodipine. | up to 144 hours post dose
t1/2 after administration of CKD-828(Fixed Dose Combination) tablet and coadministration of corresponding dose of telmisartan and s-amlodipine. | up to 144 hours post dose
AUCinf after administration of CKD-828(Fixed Dose Combination) tablet and coadministration of corresponding dose of telmisartan and s-amlodipine. | up to 144 hours post dose
Number of participants with adverse events | up to 59days post dose
  - Adverse Event monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Young-Ran Yoon, Principal Investigator — Kyungpook National University Hospital Clinical Trial Center
Locations (1):
- Kyungpook National University Hospital, Daegu, Samdeok-dong, 2-ga 50, Samdeok-dong, 2-ga 50 Jung-gu, South Korea